CLINICAL TRIAL: NCT01472536
Title: A Randomized Study of Exclusion Criteria in a University Population
Brief Title: A Study of Exclusion Criteria in a University Population
Acronym: eX-FLU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Allison Aiello, Associate Professor, Epidemiology, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 1U01CK000185-01 (NIH)
Record Dates: First submitted 2011-11-11; First posted 2011-11-16 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Influenza
Keywords: Influenza; Non pharmaceutical intervention; Sequestration; Social network
MeSH Terms: conditions — Influenza, Human | interventions — Carbon Sequestration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 3-day sequestration (Experimental): Students will be sequestered within their residence hall room for 3 days following influenza like illness symptoms
  Interventions: Behavioral: Sequestration
- Control (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Sequestration — Students will be sequestered within their residence hall room for 3 days following influenza like illness symptoms.
  Arms: 3-day sequestration

SUMMARY:
Much of community transmission of seasonal and pandemic influenza occurs in younger individuals, because of their susceptibility and their social interaction patterns.Universities are places where transmission of influenza is facilitated because of the age of individuals involved, their close contact with each other, and low vaccination coverage. Staying home when you are sick (i.e., voluntary sequestration) has been identified as one of the most efficient ways to reduce influenza transmission, but there are still insufficient data on the effects of social distancing to be able to make recommendations for future pandemics or even outbreaks of seasonal influenza.

The investigators are conducting a study on the effect of voluntary sequestration during illness on the transmission of influenza among social networks in University residence housing units at the University of Michigan. The sequestration interventions will be carried out during a period of influenza transmission that is defined by surveillance conducted at the University Health Service. Data will be collected on use of the interventions and the occurrence of influenza and other illnesses. In all selected residence halls, specimens will be collected when illness meeting a case definition for influenza-like illness occurs.

This study in a university population will evaluate the acceptability and magnitude of effect that can be expected from such an intervention, and determine the number of days that sequestration should be practiced.

ELIGIBILITY:
Inclusion Criteria:

* Live in a participating residence hall at the time of enrollment
* Be at least 18 years of age
* Be willing to report social habits and illness information electronically on a weekly basis
* Be willing to have a throat swab specimen collected if you have signs of illness during the influenza season
* Be willing to nominate close social contacts living in eligible residence halls for participation in the study
* Be willing to participate in a 3-day sequestration protocol as randomly assigned.

Exclusion Criteria:

* Non-residence in selected Residence Halls
* Unwillingness to participate in voluntary sequestration protocol and complete online surveys
* Already study employee

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1400 (Actual)
Dates: Start 2011-11; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Laboratory confirmed cases of Influenza | 10 weeks

SECONDARY OUTCOMES:
Cases of influenza like illness | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Allison E Aiello, PhD, Principal Investigator — University of Michigan; Arnold S Monto, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States